CLINICAL TRIAL: NCT01150383
Title: The Effect of Supplemental Oxygen During Physical Exercise Training on Exercise Capacity in COPD Patients.
Brief Title: SCOPE-Study: Salzburg Chronic Obstructive Pulmonary Disease- Exercise and Oxygen Study
Acronym: SCOPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Prim. Prof. MD, PhD, MBA, Paracelsus Medical University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UISM-4
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Lung Diseases, Obstructive; Respiratory Tract Diseases; Lung Diseases; Respiration Disorders; Pulmonary Disease, Chronic Obstructive; COPD; Chronic Obstructive Lung Disease; Chronic Obstructive Airway Disease; Chronic Airflow Obstruction; oxygen; oxygen supplementation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Respiratory Tract Diseases; Lung Diseases; Respiration Disorders | interventions — Physical Conditioning, Human; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group RO (Room air / Oxygen) (Active Comparator): RO (Room air / Oxygen): First 6 weeks of exercise training under normoxic conditions (Room air), followed by 6 weeks of exercise training with oxygen supplementation.
  Interventions: Other: Physical exercise training with "room air supplementation"
- group OR (Oxygen / Room air) (Active Comparator): OR (Oxygen / Room air): First 6 weeks of exercise training with oxygen supplementation, followed by 6 weeks of exercise training under normoxic conditions (room air).
  Interventions: Other: Physical exercise training with supplemental oxygen

INTERVENTIONS:
Other: Physical exercise training with supplemental oxygen — Prior to the exercise training, an intervention-free control period with usual care is planned.
  Intervention group with oxygen supplementation: Endurance training (performed within 70-80% of the heart rate at the anaerobic threshold) as well as strength training will be performed with oxygen supplementation.
  After 6 weeks of intervention with oxygen supplementation, second intervention period will start with room air instead of oxygen supplementation (as described above).
  Other Names: training; physical training; exercise
  Arms: group OR (Oxygen / Room air)
Other: Physical exercise training with "room air supplementation" — Prior to the exercise training, an intervention-free control period with usual care is planned.
  Intervention group with room air supplementation: Endurance training (performed within 70-80% of the heart rate at the anaerobic threshold) as well as strength training will be performed under normoxic conditions.
  After 6 weeks of intervention with room air, second intervention period will start with oxygen supplementation instead of room air (as described above).
  Other Names: training; physical training; exercise
  Arms: group RO (Room air / Oxygen)

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is number four of the leading causes of death in the USA and Europe. Moreover, among the top five causes of death, this disease is the only one with increasing mortality rates. Physical training has become an evidence based therapeutic intervention in these patients.

In this study the investigators aim to establish if supplemental oxygen during strength and endurance training improves exercise tolerance. Furthermore, the investigators want to research, if supplemental oxygen has the ability to increase training intensity, which would lead to a greater training effect with respect to respiratory, vascular, inflammatory and anthropometric parameters, as well as quality of life.

SCOPE is a prospective, randomized, double-blinded, controlled, cross-over trial. The investigators aim to enroll 40 patients suffering from COPD aged >30 years. Inclusion criteria are FEV1 30-60%, and PO2 at rest >55 mmHg. At baseline, patients will undergo pre-tests including pulmonary, exercise physiological and medical investigations. Prior to the exercise training, an intervention-free control period with usual care is planned. This will be followed by 2 x 6 weeks with physical training (ergometer based endurance training and strength training, using weight lifting machines) with either supplemental oxygen or usual room air (e.g.: first 6 weeks of exercise with oxygen supplementation followed by 6 weeks of room air). After the initial control period and between these two exercise periods, patients will be tested as described in pre-tests, and at the end of the second exercise training period. In addition, the investigators will assess changes in lung function and symptomatic dyspnoea, as well as in quality of life (St. George's Respiratory Questionnaire).

Within this study, the investigators hope to improve rehabilitation programs for COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* COPD with FEV1 pred. 30 to 60%, PO2 at rest > 55 mmHg and PCO2 < 45 mm Hg
* age: > 30 years

Exclusion Criteria:

* Musculoskeletal disease, which prohibits training
* Relevant neoplastic disease with cachexia
* Expected non compliance with the study protocol due to drug and alcohol abuse
* Coronary heart disease defined by angina pectoris or relevant ST-changes during exercise or myocardial infarction in the last 6 months
* Left ventricular ejection fraction < 40 %
* Renal insufficiency with creatinine > 2 mmol/liter
* Symptomatic intermittent claudication or peripheral neuropathy
* Anaemia < 10 mg/dl or red blood count < 3 Mio/mm3

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Exercise capacity (Watts/kg) | 6 weeks
  To investigate the effectiveness of physical training in COPD- patients comparing a 6 week period of exercise under oxygen supplementation with a 6 week period of exercise under "room air supplementation".

SECONDARY OUTCOMES:
Quality of life | 6 weeks
  Measured by St. George Respiratory Questionnaire
Maximal oxygen uptake (VO2-max) | 6 weeks
  Measurement of spiroergometry
Heart rate, blood pressure and exercise capacity at lactate-thresholds 2,3 and 4. | 6 weeks
  Measurement of ergometry
BODE-index | 6 weeks
  The BODE index is a simple multidimensional grading system for COPD-patients which considers body-mass index, degree of airflow obstruction (FEV1) and dyspnea (BORG scale), and exercise capacity, which will be measured by the six-minute-walk test.
Walking capacity | 6 weeks
  6-minute-walk test
Dyspnea | 6 weeks
  Measured by BORG-scale
Body composition | 6 weeks
  Body composition/muscle volume will be measured using magnetic resonance imaging.
Blood parameters of inflammation | 6 weeks
  Inflammatory changes will be assessed via blood test analysis.
Vascular changes | 6 weeks
  Vascular changes will be assessed via blood test analysis as well as analysis of endothelial function.
ten repetition maximum | 6 weeks
  The ten repetition maximum (10-RM) is a measure of the maximal weight a subject can lift 10 times.

CONTACTS AND LOCATIONS:
Overall Officials: Josef Niebauer, MD, PhD, MBA, Study Chair — Institute of Sports Medicine, Prevention and Rehabilitation, Paracelsus Medical University Salzburg
Locations (1):
- Institute of Sports Medicine, Prevention and Rehabilitation, Paracelsus Medical University Salzburg, Salzburg, Austria

REFERENCES:
- [Background] Vogiatzis I, Athanasopoulos D, Stratakos G, Garagouni C, Koutsoukou A, Boushel R, Roussos C, Zakynthinos S. Exercise-induced skeletal muscle deoxygenation in O-supplemented COPD patients. Scand J Med Sci Sports. 2009 Jun;19(3):364-72. doi: 10.1111/j.1600-0838.2008.00808.x. Epub 2009 May 19. PMID 18492053
- [Background] Nonoyama ML, Brooks D, Lacasse Y, Guyatt GH, Goldstein RS. Oxygen therapy during exercise training in chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD005372. doi: 10.1002/14651858.CD005372.pub2. PMID 17443585
- [Background] ZuWallack RL. The roles of bronchodilators, supplemental oxygen, and ventilatory assistance in the pulmonary rehabilitation of patients with chronic obstructive pulmonary disease. Respir Care. 2008 Sep;53(9):1190-5. PMID 18718038
- [Background] Watz H, Waschki B, Meyer T, Magnussen H. Physical activity in patients with COPD. Eur Respir J. 2009 Feb;33(2):262-72. doi: 10.1183/09031936.00024608. Epub 2008 Nov 14. PMID 19010994
- [Background] Puhan MA, Schunemann HJ, Frey M, Scharplatz M, Bachmann LM. How should COPD patients exercise during respiratory rehabilitation? Comparison of exercise modalities and intensities to treat skeletal muscle dysfunction. Thorax. 2005 May;60(5):367-75. doi: 10.1136/thx.2004.033274. PMID 15860711
- [Background] Casaburi R, ZuWallack R. Pulmonary rehabilitation for management of chronic obstructive pulmonary disease. N Engl J Med. 2009 Mar 26;360(13):1329-35. doi: 10.1056/NEJMct0804632. No abstract available. PMID 19321869
- [Derived] Neunhauserer D, Hudelmaier M, Niederseer D, Vecchiato M, Wirth W, Steidle-Kloc E, Kaiser B, Lamprecht B, Ermolao A, Studnicka M, Niebauer J. The Impact of Exercise Training and Supplemental Oxygen on Peripheral Muscles in Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial. Med Sci Sports Exerc. 2023 Dec 1;55(12):2123-2131. doi: 10.1249/MSS.0000000000003268. Epub 2023 Aug 2. PMID 37535316
- See also: Related Info — http://www.nlm.nih.gov/medlineplus/copdchronicobstructivepulmonarydisease.html
- See also: Related Info — http://www.salk.at/